CLINICAL TRIAL: NCT03123094
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Intravenous Dose and Single Subcutaneous Dose of BI 655130 in Healthy Japanese Male Volunteers (Double-blind, Randomised, Placebo-controlled Design).
Brief Title: Single Rising Dose Trial of Spesolimab (BI 655130) for Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1368-0009
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — spesolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Spesolimab low dose group (intravenous) (Experimental)
  Interventions: Drug: Spesolimab
- Spesolimab medium dose group (intravenous) (Experimental)
  Interventions: Drug: Spesolimab
- Spesolimab high dose group (intravenous) (Experimental)
  Interventions: Drug: Spesolimab
- Spesolimab low dose group (subcutaneous) (Experimental)
  Interventions: Drug: Spesolimab
- Placebo matching to spesolimab (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spesolimab — single dose
  Other Names: BI 655130
  Arms: Spesolimab high dose group (intravenous); Spesolimab low dose group (intravenous); Spesolimab low dose group (subcutaneous); Spesolimab medium dose group (intravenous)
Drug: Placebo — single dose
  Arms: Placebo matching to spesolimab

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of spesolimab following administration of single rising intravenous doses and single subcutaneous dose in healthy Japanese male volunteers.

Secondary objective is the exploration of the pharmacokinetics including dose proportionality of spesolimab in healthy Japanese male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood Pressure [BP], Pulse Rate [PR]), 12-lead Electrocardiogram [ECG], and clinical laboratory tests.
* Japanese ethnicity, according to the following criteria:

  -- born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who were all born in Japan
* Age of 20 to 45 years (incl.)
* Body Mass Index [BMI] of 18.5 to 25.0 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Male subjects who agree to minimize the risk of female partners being pregnant by fulfilling any of the following criteria starting from the first administration of trial medication and until 30 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom:

combined oral contraceptives, intrauterine device

* A vasectomised sexual partner (vasectomy at least 1 year prior to enrolment)
* Surgically sterilised (including hysterectomy) female partner

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure [BP], Pulse Rate [PR] or Electrocardiogram [ECG]) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections including active tuberculosis, HIV or viral hepatitis; QuantiFERON TB test will be performed at screening.
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 5 half-lives prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug.
* Administered live vaccine within 6 weeks prior to randomisation or Have plans for administration of live vaccines during the study period.
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms in males) or any other relevant Electrocardiogram [ECG] finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Further exclusion criteria apply

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Joseph D, Thoma C, Haeufel T, Li X. Assessment of the Pharmacokinetics and Safety of Spesolimab, a Humanised Anti-interleukin-36 Receptor Monoclonal Antibody, in Healthy Non-Japanese and Japanese Subjects: Results from Phase I Clinical Studies. Clin Pharmacokinet. 2022 Dec;61(12):1771-1787. doi: 10.1007/s40262-022-01176-5. Epub 2022 Dec 1. PMID 36451029
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a double-blind, randomised, and placebo-controlled trial of single rising intravenous (IV) doses and single subcutaneous (SC) doses of spesolimab (BI 655130) in healthy male Japanese subjects.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended specialist sites which would then ensure that all subjects met all inclusion/exclusion criteria. Subjects were not to be randomised to trial treatment if any one of the specific entry criteria were not met.
  Dose level for each arm cannot be provided because the information is a combination of both commercially sensitive confidential information as well as proprietary information.
Groups:
- Spesolimab Low Dose Group (Intravenous); Spesolimab Medium Dose Group (Intravenous); Spesolimab High Dose Group (Intravenous): Subjects were administered intravenously a single dose of solution for infusion of spesolimab in the range of 300 -1200 milligrams (mg) as 90 minutes infusion on day 1 of visit 2.
- Spesolimab Low Dose Group (Subcutaneous): Subjects were administered a single dose of solution for injection of spesolimab in the range of 300-1200 milligrams (mg) as subcutaneous injection on day 1 of visit 2.
- Placebo Matching to Spesolimab: Subjects administered placebo matching to spesolimab solution for infusion as intravenous as 90 min infusion or subcutaneous injection on day 1 of visit 2.
Period: Overall Study
Arm/Group | Spesolimab Low Dose Group (Intravenous) | Spesolimab Medium Dose Group (Intravenous) | Spesolimab High Dose Group (Intravenous) | Spesolimab Low Dose Group (Subcutaneous) | Placebo Matching to Spesolimab
Started | 6 | 6 | 6 | 6 | 8
Completed | 6 | 4 | 5 | 6 | 7
Not Completed | 0 | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): TS includes all subjects dispensed trial medication and documented to have taken at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Spesolimab Low Dose Group (Intravenous) | Spesolimab Medium Dose Group (Intravenous) | Spesolimab High Dose Group (Intravenous) | Spesolimab Low Dose Group (Subcutaneous) | Placebo Matching to Spesolimab | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.5 (4.51) | 31.5 (4.85) | 36.7 (3.56) | 34.7 (5.24) | 31.4 (7.65) | 33.0 (5.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 8 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 6 | 6 | 8 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug-related Adverse Events (AEs)
Description: The primary endpoint is to assess safety and tolerability of spesolimab as the number [N] of subjects with drug-related AEs.
Time Frame: From first drug administration until the end of trial examination, up to 151 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Spesolimab Low Dose Group (Intravenous) | Spesolimab Medium Dose Group (Intravenous) | Spesolimab High Dose Group (Intravenous) | Spesolimab Low Dose Group (Subcutaneous) | Placebo Matching to Spesolimab
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
Participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Area Under the Concentration-time Curve of Spesolimab in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: AUC0-∞, Area under the concentration-time curve of spesolimab in plasma over the time interval from 0 extrapolated to infinity is presented.
  Pharmacokinetic samples were collected within 2 hours pre-dose and at 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2184, 2856 and 3528 hours after dosing of dose groups with intravenous administration of spesolimab.
  Pharmacokinetic samples were collected within 2 hours pre-dose and at 0.5, 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2184, 2856 and 3528 hours after dosing of dose groups with subcutaneous administration of spesolimab.
Time Frame: Up to 3528 hours after administration of spesolimab.
Population: Pharmacokinetic (PK) set (PKS): PKS includes all subjects in the treated set who provided at least one PK parameter not excluded due to a protocol violation relevant to the evaluation of PK. Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day*microgram/millilitre [day∙μg/mL]
Arm/Group | Spesolimab Low Dose Group (Intravenous) | Spesolimab Medium Dose Group (Intravenous) | Spesolimab High Dose Group (Intravenous) | Spesolimab Low Dose Group (Subcutaneous)
Number analyzed (Participants) | 6 | 5 | 5 | 6
Day*microgram/millilitre [day∙μg/mL] | 1890 (19.9) | 3930 (18.4) | 7060 (18.0) | 1390 (24.8)
Statistical Analysis 1: Comparison: Spesolimab Low Dose Group (Intravenous) vs Spesolimab Medium Dose Group (Intravenous) vs Spesolimab High Dose Group (Intravenous); Dose proportionality was explored using the power model. Dose proportionality of spesolimab was to be assessed based on the exposure parameter AUC0-∞, determined for the 3 intravenous dose levels (perfect dose proportionality would correspond to a slope of 1); Test type: Other; Slope = 0.9533, 95% CI 2-sided [0.7810 to 1.1256], Standard Error of Mean 0.0803 — Standard error of mean is actually standard error of slope

3. Secondary Outcome: Maximum Measured Concentration of Spesolimab in Plasma (Cmax)
Description: Cmax, maximum measured concentration of spesolimab in plasma is presented. Pharmacokinetic samples were collected within 2 hours pre-dose and at 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2184, 2856 and 3528 hours after dosing of dose groups with intravenous administration of Up to 3528 hours after administration of spesolimab.
  Pharmacokinetic samples were collected within 2 hours pre-dose and at 0.5, 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2184, 2856 and 3528 hours after dosing of dose groups with subcutaneous administration of spesolimab.
Time Frame: Up to 3528 hours after administration of spesolimab.
Population: Pharmacokinetic (PK) set (PKS): PKS includes all subjects in the treated set who provided at least one PK parameter not excluded due to a protocol violation relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/millilitre [μg/mL]
Arm/Group | Spesolimab Low Dose Group (Intravenous) | Spesolimab Medium Dose Group (Intravenous) | Spesolimab High Dose Group (Intravenous) | Spesolimab Low Dose Group (Subcutaneous)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Microgram/millilitre [μg/mL] | 99.7 (10.4) | 193.0 (17.9) | 400.0 (12.9) | 32.2 (21.8)
Statistical Analysis 1: Comparison: Spesolimab Low Dose Group (Intravenous) vs Spesolimab Medium Dose Group (Intravenous) vs Spesolimab High Dose Group (Intravenous); Dose proportionality was explored using the power model. Dose proportionality of spesolimab was to be assessed based on the exposure parameter Cmax, determined for the 3 intravenous dose levels (perfect dose proportionality would correspond to a slope of 1); Test type: Other; Slope = 1.0014, 95% CI 2-sided [0.8809 to 1.1219], Standard Error of Mean 0.0568 — Standard error of mean is actually standard error of slope

4. Secondary Outcome: Total Clearance of Spesolimab in Plasma After Intravenous Administration (CL)
Description: CL, total clearance of spesolimab in plasma after intravenous administration is presented for intravenous dose groups.
Time Frame: Pharmacokinetic samples were collected within 2 hours (h) pre-dose and at 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, 168, 336, 504, 672, 840, 1008, 1344, 1680, 2184, 2856 and 3528 h after dosing of dose groups with intravenous administration of spesolimab.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre/day [L/day]
Arm/Group | Spesolimab Low Dose Group (Intravenous) | Spesolimab Medium Dose Group (Intravenous) | Spesolimab High Dose Group (Intravenous)
Number analyzed (Participants) | 6 | 5 | 5
Litre/day [L/day] | 0.159 (19.9) | 0.153 (18.4) | 0.170 (18.0)

5. Secondary Outcome: Volume of Distribution at Steady State After Intravenous Administration of Spesolimab (Vss)
Description: Vss, volume of distribution at steady state after intravenous administration of spesolimab is presented for intravenous dose groups.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre [L]
Arm/Group | Spesolimab Low Dose Group (Intravenous) | Spesolimab Medium Dose Group (Intravenous) | Spesolimab High Dose Group (Intravenous)
Number analyzed (Participants) | 6 | 5 | 5
Litre [L] | 6.19 (18.1) | 6.97 (11.9) | 6.60 (11.6)

ADVERSE EVENTS:
Time Frame: From first drug administration until the end of trial examination, up to 151 days.
Description: Treated set (TS): TS includes all subjects dispensed trial medication and documented to have taken at least one dose of investigational treatment.
Groups:
- Spesolimab High Dose Group: Subjects administered single dose of 1200 mg BI 655130 solution for infusion as intravenous as 90 min infusion on day 1 visit 2.
Arm/Group | Spesolimab Low Dose Group (Intravenous) | Spesolimab Medium Dose Group (Intravenous) | Spesolimab High Dose Group | Spesolimab Low Dose Group (Subcutaneous) | Placebo Matching to Spesolimab
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 1/6 | 0/6 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Spesolimab Low Dose Group (Intravenous) (N=6) | Spesolimab Medium Dose Group (Intravenous) (N=6) | Spesolimab High Dose Group (N=6) | Spesolimab Low Dose Group (Subcutaneous) (N=6) | Placebo Matching to Spesolimab (N=8)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT03123094/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT03123094/SAP_001.pdf